CLINICAL TRIAL: NCT02934854
Title: Biomarker for Creatine Deficiency Syndromes. An International, Multicenter, Epidemiological Study.
Brief Title: Biomarker for Creatine Deficiency Syndromes (BioCDS)
Acronym: BioCDS
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BCDS 06-2018
Record Dates: First submitted 2016-09-19; First posted 2016-10-17 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Intellectual Disability; Developmental Delay; Movement Disorder; Behavioral Disorder; Intractable Epilepsy
Keywords: Creatine Transporter Deficiency (CTD); Guanidinoacetate Methyltransferase Deficiency (GAMT); Arginine: Glycine Amidinotransferase Deficiency (AGAT); Biomarker
MeSH Terms: conditions — Intellectual Disability; Learning Disabilities; Movement Disorders; Mental Disorders; Drug Resistant Epilepsy; Creatine deficiency, X-linked; Guanidinoacetate methyltransferase deficiency; Arginine-Glycine Amidinotransferase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, maximal 7,5 ml of blood will be taken via using a dry blood spot filter card. To proof the correct Creatine Deficiency Syndromes diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Creatine Deficiency Syndromes will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with the Creatine Deficiency Syndromes or high-grade suspicion for the Creatine Deficiency Syndromes

SUMMARY:
Development of a new mass spectrometry-based biomarker for the ear-ly and sensitive diagnosis of the Creatine Deficiency Syndromes from dry-blood-spot sample

DETAILED DESCRIPTION:
The Creatine Deficiency Syndromes (CDS) are a group of inborn errors of metabolism which interrupt the biosynthesis or transportation of creatine. Individuals with CDS classically present neurological symptoms (seizures, movement disorders and myopathy), and behavioral manifestations. This group includes two creatine biosynthesis disorders (Guanidinoacetate Methyltransferase Deficiency and L-Arginine: Glycine Amidinotransferase Deficiency), as well as X-linked Creatine Transporter Deficiency.

Guanidinoacetate Methyltransferase Deficiency:

Guanidinoacetate Methyltransferase Deficiency is inherited in an autosomal recessive manner and is caused by biallelic mutations in the GAMT gene. This gene maps to 19p13.3 and is involved in the biosynthesis of creatine. Individuals with this deficiency typically present with severe intellectual disabilities and seizure disorders which may be resistant to drug therapy. Behavioral problems, including autistic behaviors and self-mutilation are common, and pyramidal/extrapyramidal symptoms affect about one-half of patients. Dietary management via manipulation of critical amino acids may improve clinical outcome. Mutations in the GAMT gene are a relatively rare cause of creatine deficiency syndrome.

L-Arginine: Glycine Amidinotransferase Deficiency:

L-Arginine: Glycine Amidinotransferase Deficiency is a very rare type of CDS characterized by global developmental delay, appearing in infancy, which can be associated with language impairment and autistic behavior in some, as well as a mild to moderate intellectual disability. Progressive muscle weakness and fatigability have been reported in older patients. Seizures and failure to thrive have also been described. If creatine supplementation is administered early enough, psychomotor delay may be avoided. This deficiency is caused by mutations in GATM gene, located to chromosome 15q15.1. This gene encodes the enzyme L-Arginine: Glycine Amidinotransferase, which converts arginine and glycine to ornithine and guanidinoacetate in the creatine cycle pathway. This deficiency is transmitted in an autosomal recessive manner.

X-linked Creatine Transporter Deficiency:

X-linked Creatine Transporter Deficiency is a creatine deficiency syndrome characterized clinically by global developmental delay, intellectual disability with prominent speech/language delay, autistic behavior and seizures. Affected individuals may present low weight gain, muscular hypotonia, and poor muscle mass. Subtle dysmorphic features such as midface hypoplasia, long face, and prominent chin have been reported in various affected male patients. In adult patients, cardiac and gastrointestinal disorders have been reported. The onset of symptoms occurs during infancy, usually before the age of 2 years. Males are mainly affected, but females can also have various degrees of severity of disease manifestations. This deficiency has been reported in more than 150 individuals worldwide and is mostly due to frameshift and splicing mutations in the creatine transporter gene SLC6A8 (Xp28).

New methods, like mass-spectrometry, give a good chance to characterize specific metabolic alterations in the blood of affected patients, that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of the Creatine Deficiency Syndromes or a high-grade suspicion for the Creatine Deficiency Syndromes

High-grade suspicion is present, if one or more inclusion criteria are valid:

* Positive family anamnesis for the Creatine Deficiency Syndromes
* Intellectual disability
* Seizure disorder of variable severity
* Developmental delay
* Speech/language delay
* Movement disorder
* Behavioral disorder (autism, hyperactivity, self-injury)
* Intractable epilepsy

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Creatine Deficiency Syndromes or no valid criteria for profound suspicion of the Creatine Deficiency Syndromes

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the Creatine Deficiency Syndromes or high-grade suspicion for the Creatine Deficiency Syndromes
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Creatine Deficiency Syndromes related genes | 4 weeks
  Next-Generation Sequencing (NGS) of the genes SLC6A8, GAMT, and GATM will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Creatine Deficiency Syndromes specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Egypt (2):
  - Ain Shams University, Medical Genetics Center, Cairo
  - Chindren's hospital, Faculty of Medicine, Ain Shams University, Cairo
- Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided